CLINICAL TRIAL: NCT01612806
Title: A Multi-center, Prospective, Randomized Study With PriMatrix Dermal Repair Scaffold, PriMatrix Ag Antimicrobial Dermal Repair Scaffold, and Standard of Care for the Treatment of Venous Leg Ulcers
Brief Title: A Multi-center, Prospective, Randomized Study With PriMatrix and PriMatrix Ag for the Treatment of Venous Leg Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Site selection
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEI-006
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Venous Stasis Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PriMatrix (Experimental): PriMatrix Dermal Repair Scaffold
  Interventions: Device: PriMatrix; Procedure: moist wound therapy
- PriMatrix Ag (Experimental): PriMatrix Ag Antimicrobial Dermal Repair Scaffold
  Interventions: Device: PriMatrix Ag; Procedure: moist wound therapy
- Standard of Care (Active Comparator): Standard of Care Moist Wound Therapy
  Interventions: Procedure: moist wound therapy

INTERVENTIONS:
Device: PriMatrix — fetal bovine dermal scaffold
  Arms: PriMatrix
Device: PriMatrix Ag — fetal bovine dermal scaffold with Ag
  Arms: PriMatrix Ag
Procedure: moist wound therapy — standard of care moist wound therapy

SUMMARY:
To evaluate the effectiveness of PriMatrix, PriMatrix Ag, and Standard of Care in the treatment of venous leg ulcers (VLUs).

DETAILED DESCRIPTION:
Healing percentages

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age
* Ankle-brachial index (ABI) > 0.80
* Study wound 2-64 cm2 surface area
* Wound does not exhibit a greater than 50% reduction in surface area during the screening period

Exclusion Criteria:

* Suspected or confirmed signs/symptoms of wound infection
* Hypersensitivity to bovine collagen
* Body Mass Index (BMI) ≥ 45

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Percent of VLUs healed by week 12 post-randomization | 12 weeks

SECONDARY OUTCOMES:
Cost of treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Starinski, DPM, Study Director — TEI
Locations (5):
- Puerto Rico (5):
  - Caribbean Clinical Trials, San Juan, PR
  - Dr. Pila Metropolitan Hospital Wound Healing Center, Ponce
  - Doctors' Center Hospital of San Juan, San Juan
  - Wound and Ulcer Care Clinic of San Juan, San Juan
  - Wilma N. Vazquez Hospital, Vega Baja